CLINICAL TRIAL: NCT01060566
Title: An Open-Label Phase 1 Study to Examine the Effect of VX-770 on Midazolam and Rosiglitazone and the Effect of Fluconazole on VX-770 in Healthy Subjects
Brief Title: Study of VX-770 on Midazolam and Rosiglitazone and the Effect of Fluconazole on VX-770
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Medical Monitor, Vertex Pharmaceuticals Incorporated
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX09-770-010
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- VX-770 (Experimental)
  Interventions: Drug: VX-770
- Midazolam (Experimental)
  Interventions: Drug: VX-770
- Rosiglitazone (Experimental)
  Interventions: Drug: VX-770
- Fluconazole (Experimental)
  Interventions: Drug: VX-770

INTERVENTIONS:
Drug: VX-770 — In period 1, subjects will receive a single oral dose of midazolam (2 mg) and on Day 1 and Day 8. Subjects will receive single oral dose of rosiglitazone 4 mg and on Day2 and Day 9. Subjects will receive multiple doses of VX-770 150 mg q12h Day 3-10.
  Arms: Midazolam; Rosiglitazone; VX-770
Drug: VX-770 — In period 2, subjects will receive 150 mg VX-770 q12h orally from Day 1 through the morning of Day 8. On the morning of Period 2 Day 1, subjects will receive a 400 mg loading dose of fluconazole. Thereafter, subjects will receive 200 mg fluconazole qd orally from Day 2 through Day 9.
  Arms: Fluconazole; VX-770

SUMMARY:
The objectives of this study are to evaluate the effects of VX-770 on Midazolam and Rosiglitazone, and the effect of Fluconazole on VX-770.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male or female and between 18 and 55 years of age.
* Subjects must be judged to be in good health.
* Subjects must have a body mass index (BMI) from 18 to 30 kg/m2.

Exclusion Criteria:

* History of any illness that, in the opinion of the investigator or the subject's general practitioner, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject.
* Subjects who have human immunodeficiency virus (HIV), hepatitis C, or active hepatitis B.
* Female subjects and female partner(s) of male subjects who are pregnant, nursing, or planning to become pregnant during the study or within 90 days of the last dose of study drug.
* History of cardiovascular disease, hypoglycemia, or edema.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Midazolam, Rosiglitazone and VX 770 pharmacokinetic (PK) parameter | 11 days
Fluconazole and VX 770 PK parameters | 10 days

SECONDARY OUTCOMES:
1´ hydroxy midazolam PK parameters in plasma | 11 days
Safety as measured by adverse events, physical examinations, vital signs, ECGs, and clinically significant laboratory assessments | 21 days
Metabolites PK parameters in plasma | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: H. Frank Farmer, MD, Principal Investigator — Covance CRU, Inc.
Locations (1):
- Covan CRU, Inc., Daytona Beach, Florida, United States